CLINICAL TRIAL: NCT01339897
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study Evaluating the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of N6022 in Healthy Subjects
Brief Title: A Safety Study Evaluating N6022 in Multiple-Ascending Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N6022-1H1-03
Record Dates: First submitted 2011-04-19; First posted 2011-04-21 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: N6022, GSNORi
MeSH Terms: interventions — N6022; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 5 mg/N6022 (Active Comparator): Injectable formulation, given at doses per cohort of 5 mg given QD each day over 7 days.
  Interventions: Drug: 5 mg/N6022
- Placebo (Placebo Comparator): Injectable formulation normal saline
  Interventions: Drug: Placebo
- 10mg/N6022 (Active Comparator): Injectable formulation, given at doses of 10 mg given QD each day over 7 days.
  Interventions: Drug: 10mg/N6022
- 20mg/N6022 (Active Comparator): Injectable formulation, given at doses per cohort of 20 mg given QD each day over 7 days.
  Interventions: Drug: 20mg/N6022

INTERVENTIONS:
Drug: 5 mg/N6022 — Intravenous formulation, given at doses of 5 mg once each day over 7 days.
  Other Names: N6022; GSNOR Inhibitor
  Arms: 5 mg/N6022
Drug: Placebo — Same administration procedures as active
  Other Names: Normal Saline
  Arms: Placebo
Drug: 10mg/N6022 — Intravenous formulation given at doses of 10 mg once each day over 7 days.
  Other Names: N6022; GSNOR Inhibitor
  Arms: 10mg/N6022
Drug: 20mg/N6022 — Intravenous formulation given at doses of 20 mg once each day over 7 days.
  Other Names: N6022; GSNOR Inhibitor
  Arms: 20mg/N6022

SUMMARY:
This Phase 1 study will evaluate multiple doses across a range that has been found to be effective in mouse models of asthma and safe in one Phase 1 clinical trial. It is intended to provide evidence of the tolerability of multiple doses as well as provide information on the Pharmacokinetic (PK) and metabolism of N6022 in humans.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multiple ascending dose study, in at least three ascending cohorts. Twenty-four subjects will be enrolled initially in the first three cohorts, with up to 40 subjects to be enrolled overall if additional cohorts are required to reach the maximum tolerated dose (MTD). The cohorts will be enrolled in two groups of 4 each with approximately 7 days between groups to conduct safety monitoring committee review for approval to proceed to the second group in the cohort. Eight subjects will be enrolled per cohort, randomized 3:1 to N6022: placebo. Each subject will undergo screening (Day -28 to Day -2) and, if eligible, they will be instructed to begin a low-nitrate diet on Day -4. Subjects will return to the clinical site on Day -1, and eligibility will be reconfirmed. Eligible subjects will receive a dose of investigational medicinal product ([IMP], N6022 or placebo) by intravenous (IV) infusion on study Days 1 through 7 and will be followed for safety, PK, and PD until discharge on the morning of Day 8. Subjects will return to the clinic for a follow-up visit on Day 15 (± 1 day) and will be contacted via telephone on Day 28 (± 1 day) for the end-of-study safety follow-up visit. Participation of an individual subject may last approximately 56 days from the time of screening until the end-of-study follow-up visit.

A Safety Monitoring Committee (SMC) will review the safety data in each cohort after the Day 15 Follow-up visit, before proceeding to the next ascending dose cohort, modifying the dose, repeating a dose, or stopping the study according to the stopping rules outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is healthy, determined by pre-study medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations
2. Subject is a non-smoker (or other nicotine user) as determined by history (no nicotine use over the past year) and a negative urine cotinine test at screening and Day 1.
3. Subject has a body weight > 50 kg and BMI between 19.5 and 29.5 kg/m2, inclusive, at screening.
4. Subject has systolic BP > 90 mmHg and diastolic BP > 50 mmHg at screening or Day-1.

Exclusion Criteria:

1. Subject has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the investigator or designee.
2. Subject is a current alcohol abuser and/or has a history of illicit drug abuse within six months of entry.
3. Subject has donated blood (> 500 mL) or blood products within 56 days prior to Day -1.
4. Subject has a history of bleeding disorders (i.e., severe hemorrhage, melena, rectal bleeding, nosebleeds, bruising, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MDCM, MSc(A), Principal Investigator — Parexel
Locations (1):
- Parexel International, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 06April2011 and 09August2011. This study was done at a single Phase 1 site.
Groups:
- 5 mg/N6022: Active Group- 5 mg by IV administration (5 mg/minute)
- Placebo: Non-Active
- 10 mg/N6022: Active Group- 10 mg by IV administration (5 mg/minute)
- 20 mg/N6022: Active Group- 20 mg by IV administration (5 mg/minute)
Period: Overall Study
Arm/Group | 5 mg/N6022 | Placebo | 10 mg/N6022 | 20 mg/N6022
Started | 7 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received any amount of IMP
Groups:
- Cohort 1: N6022 - Active 5 mg
- Cohort 2: N6022 - Active 10 mg
- Cohort 3: N6022 - Active 20 mg
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 6 | 6 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 32 [25 to 39] | 31 [22 to 45] | 35 [22 to 45] | 35 [25 to 45] | 33 [22 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 6 | 6 | 6 | 25
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 6 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety of Escalating Multiple Doses of N6022 in Healthy Subjects
Description: Safety variables (adverse events, vital signs, physical examination, telemetry, 12-lead ECG, infusion site reactions, O2 saturation, and clinical laboratory assessments)
Time Frame: Over 7 days
Population: Any subject that received any dose of N6022 or placebo.
Measure: Number; unit: participants
Groups:
- Cohort 2: N6022 Active - 10 mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6
participants
  Number of subjects on study | 7 | 6 | 6 | 6
  Early Termination | 1 | 0 | 1 | 0
  Treatment related AE | 0 | 0 | 1 | 0

2. Secondary Outcome: Pharmacokinetics of N6022
Description: N6022 AUC0-tau measurements from Day 1
Time Frame: Day 1, 24 hours
Population: Any subject that completed N6022 or placebo PK sampling
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Cohort 1: N6022 Active - 5 mg
- Cohort 3: N6022 Active - 20 mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6
h*ng/mL | 138 (13.0) | 334 (21.1) | 669 (16.9) | 0 (0)

3. Secondary Outcome: Pharmacokinetics of N6022 Over 7 Days
Description: Analysis of N6022 AUC0-tau values from Study Day 7
Time Frame: Day 7, 24 hours
Population: N6022 AUC0-tau values from Study Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6
h*ng/mL | 149 (24.6) | 367 (14.2) | 811 (11.3) | 0 (0)

4. Secondary Outcome: Pharmacokinetics of N6022 on Study Day 1
Description: Analysis of N6022 Cmax values on Study Day 1
Time Frame: Day 1, 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6
ng/mL | 465 (69.8) | 1270 (95.6) | 1400 (86.2) | 0 (0)

5. Secondary Outcome: Pharmacokinetics of N6022 Cmax Values on Study Day 7
Description: Pharmacokinetic Analysis of N6022 Cmax values on Study Day 7
Time Frame: Day 7, 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6
ng/mL | 287 (89.8) | 1110 (34.1) | 2320 (13.5) | 0 (0)

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 2/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=6) | Cohort 3 (N=6) | Placebo (N=6)
Ventricular Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Isolated episode, non-sustained
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — administration and site conditions
Injection Site Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — administration and site conditions
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — administration and site conditions
Otitis Externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculosketetal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — administration and site conditions
Upper Respiratory tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Magnesium Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pre-syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — administration and site conditions
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — administration and site conditions
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Phlebitis Superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the investigator's name, address, qualifications, and extent of involvement. An investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted with the Sponsor in advance.